CLINICAL TRIAL: NCT05014594
Title: Sodium-glucose Linked Transporter 2 (SGLT-2) Inhibitors in Recurrent Ascites: a Pilot RCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr.Virendra Singh, Professor and Head, Department of Hepatology, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dapa recurrent ascites
Record Dates: First submitted 2021-08-14; First posted 2021-08-20 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Cirrhosis; Ascites Hepatic
MeSH Terms: conditions — Fibrosis | interventions — dapagliflozin; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Dapaglifozin) (Active Comparator): Group A will receive oral Dapaglifozin (10 mg/day) along with standard medical therapy for 6 months
  Interventions: Drug: Dapagliflozin (10Mg Tab) along with standard medical therapy
- Group B (Placebo) (Placebo Comparator): Group B will receive placebo of Dapaglifozin along with standard medical therapy for 6 months
  Interventions: Drug: Placebo of dapaglifozin along with standard medical therapy

INTERVENTIONS:
Drug: Dapagliflozin (10Mg Tab) along with standard medical therapy — Oral Dapaglifozin (10 mg/day) along with standard medical therapy will be given to Group A while a placebo of dapaglifozin along with standard medical therapy will be used in Group B
  Arms: Group A (Dapaglifozin)
Drug: Placebo of dapaglifozin along with standard medical therapy — Standard medical therapy will include dietary restriction of sodium, treatment with diuretics, repeated LVP as needed and other supportive care. Patients on non-selective beta blockers will continue to do so with dose modifications/withdrawal as per Baveno VI guidelines.
  Arms: Group B (Placebo)

SUMMARY:
The development of ascites is a landmark event in the natural history of cirrhosis and signifies a grim prognosis. Portal hypertension and splanchnic arterial vasodilatation are the major contributors in the development of ascites. Vasodilatation with the consequential decrease in effective circulating volume leads to the activation of sympathetic nervous system and renin angiotensin aldosterone system (RAAS), leading to antinatriuretic effects and retention of sodium and water. This results in the formation of ascites. Management of ascites primarily consists of salt restrictrion and diuretics. Liver transplant is the ultimate panacea.

Dapaglifozin, a Sodium glucose linked transporter-2(SGLT-2) inhibitor, is a part of the routine armamentarium for treatment of patients with Diabetes Mellitus type-2. Its safety is well established in non-diabetic patients too where it has been shown to improve cardiovascular outcomes. The risk of hypoglycemia is negligible as its action is independent of insulin. By virtue of its natriuretic effect, it has been shown to reduce hospitalisations in patients with heart failure irrespective of the presence of diabetes. We hypothesise that a similar natriuretic effect may help in suppressing the renin-angiotensin axis with improved mobilization of ascites in patients with cirrhosis. Pharmacokinetic data on the use of Dapaglifozin suggest that there is no need for dose modification in cirrhosis. The AUC and Cmax for Dapaglifozin in Child Pugh C cirrhosis is 67% and 40%, respectively. In a recent small case series, SGLT-2 inhibitors including dapaglifozin led to improvement in fluid retention and serum sodium, without acute kidney injury or encephalopathy, in patients with cirrhosis. However, SGLT-2 inhibitors have not been evaluated in randomized controlled trials. In this pilot study, we plan to evaluate the efficacy and safety of dapaglifozin in cirrhotics patients with recurrent ascites.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years
2. Cirrhosis as determined by clinical findings, hemogram and liver function tests, endoscopic findings and imaging
3. Recurrent ascites: Recurrent ascites will be defined as tense ascites recurring at least thrice within the last 1-year despite optimal standard medical treatment including large volume paracentesis and diuretics

Exclusion Criteria:

1. Presence of chronic kidney disease as defined by an estimated glomerular filtration rate of <60 ml/min for more than 3 months. The MDRD-6 equation will be used for estimating GFR.
2. Portal vein thrombosis
3. Hepatocellular carcinoma.
4. Gastrointestinal bleed in the preceding 2-weeks
5. Overt hepatic encephalopathy in the preceding 1-month
6. Documented hypoglycemia in the preceding 1-month
7. Serum sodium < 125 meq/l
8. History of skeletal fracture in the preceding year or any past history of fragility fracture
9. History of peripheral vascular disease
10. Acute kidney injury as defined by the International Club of Ascites criteria
11. Infection within 1-month preceding the study
12. Anatomic urologic defects that predispose to urinary tract infection
13. Mixed ascites (additional etiology of ascites apart from portal hypertension)
14. Any severe extra hepatic condition including respiratory and cardiac failure
15. Acute-on-chronic liver failure as per the APASL or CANONIC criteria
16. Treatment with drug with known effects on systemic and renal hemodynamics within 7 days of inclusion excepting beta-blockers
17. Patients opting for liver transplant or TIPS
18. Refusal to give consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2022-05-19 (Estimated); Study Completion 2022-05-19 (Estimated)

PRIMARY OUTCOMES:
control of ascites at 6-months | 6 months
  Control of ascites will be defined as follows-
  * Complete response will be total absence of ascites.
  * Partial response as presence of ascites not requiring paracentesis
  * Non response will be defined as persistence of severe ascites requiring paracentesis.

SECONDARY OUTCOMES:
Change in eGFR measured by MDRD-6 at 3 months and 6 months | 6 months
  eGFR will be measured by MDRD-6 formula
Change in urine output at 2-weeks, 3-months and 6-months | 6-months
  Change in 24-hour urine output (ml) at 6-months
Change in serum sodium (mEq/l) at 2-weeks, 3-months and 6 months | 6 months
  Change in serum sodium (mEq/l)
Change in 24-hours urinary sodium (mEq) at 2 weeks, 3 months and 6 months | 6 months
  Change in 24-hours urinary sodium (mEq)
Change in HbA1c at 3 and 6 months | 6 months
  Change in HbA1c
Change in Child-Turcotte-Pugh (CTP) score at 3 months and 6 months | 6 months
  Change in CTP score. The CTP score incorporates the variables of serum bilirubin, albumin, prothrombin time-INR, grade of ascites and hepatic encephalopathy. The score ranges from 5-15 and a higher score portends a worse prognosis
Change in model for end stage liver disease (MELD) score at 3 months and 6 months | 6 months
  Change in MELD score. The MELD score incorporates the variables of serum bilirubin, creatinine and Internation Normalised Ratio (INR). Higher MELD score indicates worse prognosis
Incidence of spontaneous bacterial peritonitis (SBP), urinary tract infection (UTI) and other infections | 6 months
  The diagnosis of SBP will be based on neutrophil count in ascitic ﬂuid of >250/mm3 as determined by microscopy and positive ascitic fluid culture or >250 /mm3 with negative culture called as culture negative neutrocytic ascites.Other infections will be diagnosed as per CDC criteria.
Incidence of overt hepatic encephalopathy over 6-months | 6 months
  Over hepatic encephalopathy (HE) will be defined as grade II or higher HE as per the West haven classification
Incidence of acute kidney injury over 6-months | 6 months
  Acute kidney injury will be defined as per the International Club of Ascites criteria
Incidence of Hyponatremia (serum sodium <130 meq/L), hypokalemia (Serum potassium < 3.5 meq/L), hyperkalemia (Serum potassium >6meq/L) over 6-months. | 6 months
  Hyponatremia: serum sodium <130 meq/L hypokalemia: serum potassium < 3.5 meq/L hyperkalemia: serum potassium >6meq/L)
Incidence of skeletal fractures over 6-months | 6 months
  Incidence of skeletal fractures over 6-months
Change in bone densitometry as assessed by DEXA at 6-months | 6 months
  Bone densitometry will be assessed by DEXA
Incidence of diabetic ketoacidosis or hyperglycemic hyperosmolar nonketotic coma over 6-months | 6 months
  Incidence of diabetic ketoacidosis or hyperglycemic hyperosmolar nonketotic coma over 6-months
Incidence of hepatocellular carcinoma over 6-months | 6 months
  Hepatocellular carcinoma will be diagnosed based on imaging findings and AFP
Changes in plasma renin activity and aldosterone levels at 6- months | 6 months
  Changes in plasma renin activity (ng/ml/hr) and aldosterone (ng/dL) levels at 6- months
Frequency and volume of LVP over 6-months. | 6 months
  Frequency and volume of ascitic fluid removed (in litres) over 6-months.
Survival at 6-months | Survival at 6-months
  Survival at 6-months after start of therapy
Safety of dapaglifozin as assessed by adverse effects | 6 months
  Safety of dapaglifozin as assessed by adverse effects
Renal resistive index at 6 months | 6 months
  Renal resistive index will be measured using ultrasound doppler interrogation of intrarenal arteries using formula (peak systolic velocity - end-diastolic velocity) / peak systolic velocity

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Hepatology, PGIMER, Chandigarh, India

REFERENCES:
- [Derived] Singh V, De A, Aggrawal R, Singh A, Charak S, Bhagat N. Safety and Efficacy of Dapagliflozin in Recurrent Ascites: A Pilot Study. Dig Dis Sci. 2025 Feb;70(2):835-842. doi: 10.1007/s10620-024-08667-4. Epub 2024 Oct 9. PMID 39384712